CLINICAL TRIAL: NCT00777530
Title: Ascending Single-Dose Of The Safety, Tolerability, And Pharmacokinetics Of Bosutinib Administered Orally With Multiple Doses Of Ketoconazole To Healthy Adult Subjects.
Brief Title: Study Evaluating Ascending Single-Dose Of Bosutinib Administered With Multiple Doses Of Ketoconazole To Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: 3160A4-1114
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Breast Cancer; Tumors; Leukemia
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Leukemia | interventions — bosutinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Bosutinib (SKI-606)

INTERVENTIONS:
Drug: Bosutinib (SKI-606)

SUMMARY:
The purpose of this study is to assess the safety and tolerability of ascending single oral doses of bosutinib administered with multiple doses of ketoconazole and to provide the pharmacokinetic profile of bosutinib when administered with multiple doses of ketoconazole and with food in healthy adult subjects.

ELIGIBILITY:
Inclusion criteria:

1. Men or women of nonchildbearing potential (WONCBP) aged 18 to 50 years inclusive on study day 1. WONCBP may be included if they are either surgically sterile (hysterectomy and/or oophorectomy) or postmenopausal for ≥ 1 year (with follicle-stimulating hormone [FSH] ≥ 38 mIU/mL) and must have a negative serum pregnancy test result before administration of test article.
2. Body mass index (BMI) in the range of 18.0 to 30.0 kg/m2 and body weight ≥ 50 kg.
3. Healthy as determined by the investigator on the basis of screening evaluations.

Exclusion criteria:

1. Family history QT prolongation, syncope, seizure, or unexplained cardiac related death.
2. Presence or history of any disorder that may prevent the successful completion of the study.
3. Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Safety based on adverse events monitoring, physical examinations, vital sign evaluations, 12-lead ECGs and routine laboratory tests. | 5 weeks

SECONDARY OUTCOMES:
Blood samples | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Utrecht, Netherlands

REFERENCES:
- [Derived] Abbas R, Leister C, El Gaaloul M, Chalon S, Sonnichsen D. Ascending single-dose study of the safety profile, tolerability, and pharmacokinetics of bosutinib coadministered with ketoconazole to healthy adult subjects. Clin Ther. 2012 Sep;34(9):2011-9.e1. doi: 10.1016/j.clinthera.2012.07.006. Epub 2012 Aug 9. PMID 22884766